CLINICAL TRIAL: NCT07187557
Title: The Effect of Self-Compassion Based Birth Preparation Program on Self-Compassion, Body Image, Fear of Childbirth, Depression, Anxiety and Stress in Pregnant Women
Brief Title: The Effect of Self-Compassion Based Birth Preparation Program
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Hilal Gül Boyraz Yanik, Research Assistant, Ordu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 07.02.2025/34
Record Dates: First submitted 2025-06-11; First posted 2025-09-23 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Pregnant Women

STUDY DESIGN:
Intervention Model Description: There is an intervention and control group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention)
- A self-compassion based birth preparation program group (Experimental): A self-compassion based birth preparation program
  Interventions: Other: A self-compassion based birth preparation program

INTERVENTIONS:
Other: A self-compassion based birth preparation program — A self-compassion based birth preparation program
  Arms: A self-compassion based birth preparation program group

SUMMARY:
The pregnancy period, during which physiological, psychological and social changes occur, can negatively affect women mentally. It is stated that women's concerns about their own and their baby's health, anxiety and fear regarding birth, the uncertainty of the postpartum process and ambivalent feelings experienced cause negative mood changes. During pregnancy, body image dissatisfaction may develop due to weight gain, posture and skin changes, and this may cause women to experience depressive symptoms. Psychological changes such as depression, anxiety and stress experienced during pregnancy cause women to experience fear and anxiety regarding birth. Fear of birth, which is affected by many factors, also affects women's birth preferences and method. Fear of birth also affects women's psychological well-being in the postpartum period. Interventions are needed to ensure and maintain the psychological resilience of pregnant women. The aim of this study is to determine the effect of a self-compassion-based birth preparation program on self-compassion, body image, fear of birth, depression, anxiety and stress.

ELIGIBILITY:
Inclusion Criteria:

* Those who are 18 years of age and older,

  * Those who have at least primary school education,
  * Those who understand and speak Turkish,
  * Those who reside within the borders of Ordu province,
  * Those who have no obstacle to vaginal birth,
  * Those who conceive naturally,
  * Those who have a singleton pregnancy,
  * Those who are 28 weeks or more pregnant,
  * Pregnant women who agree to participate in the study will be included.

Exclusion Criteria:

* - Those who have a history of risky pregnancies,
* Those who have chronic and/or psychiatric health problems,
* Those who have a cesarean section indication will not be included in the study. Exclusion criteria for the study
* Those who are planned for a cesarean section due to medical indications at any stage of the study,
* Those who do not attend at least three sessions of the education program,
* Those who are at risk during the pregnancy at any stage of the study,
* Pregnant women who start labor while the study is ongoing will be excluded from the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-09-24 (Actual); Primary Completion 2026-06-12 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
The Effect of Self-Compassion Based Birth Preparation Program on Self-Compassion, Body Image, Fear of Childbirth, Depression, Anxiety and Stress in Pregnant Women | from june 2025 to june 2026
  This study aims to determine the effects of a self-compassion-based birth preparation program on self-compassion, body image, fear of childbirth, depression, anxiety and stress in pregnant women
Personal Information Form | In the 28th week of pregnancy
  Developed by the researchers based on literature, the form consists of questions regarding the socio-demographic and obstetric characteristics of pregnant women, such as their age, educational status, employment status, chronic disease status, number of pregnancies, gestational age, and number of children.
Self-Compassion Scale Short Form | At 28 weeks of pregnancy, after completing the program (4 weeks later) 1st month postpartum 3rd month postpartum
  The Self-Compassion Scale Short Form, developed by Raes et al. (2011), is used to measure an individual's level of self-compassion. The scale was adapted into Turkish by Yıldırım and Sarı (2018). The single-dimension scale consists of 11 items and a 5-point Likert-type scale. High scores indicate high levels of self-compassion. The lowest possible score is 11, and the highest is 55. There is no cut-off score for the scale
Pregnancy Body Image Scale | At 28 weeks of pregnancy, after completing the program (4 weeks later)
  The Pregnancy Body Image Scale was developed by Watson et al. (2017) and adapted into Turkish by Gün Kakaşçı et al. (2022). As the total score on the scale increases, the perception of negative body image in pregnant women increases. The Cronbach's alpha coefficient for the entire scale was 0.90 and ranged from 0.65 to 0.94 for its subscales
Wijma Childbirth Expectation/Experience Scale Version A | At 28 weeks of pregnancy, after completing the program (4 weeks later)
  This six-point Likert-type scale, consisting of 33 items covering childbirth-related fears, is scored from 0 to 5, with 0 being interpreted as completely and 5 being interpreted as not at all. The minimum score on the W-DEQ-A is 0, and the maximum score is 165. As women's scale scores increase, their fear of childbirth increases. W-DEQ-A scores are graded into four groups: mild fear of childbirth (W-DEQ-A score ≤37), moderate fear of childbirth (W-DEQ-A scores between 38 and 65), severe fear of childbirth (W-DEQ-A scores between 66 and 84), and clinical fear of childbirth (W-DEQ-A scores ≥85.
Wijma Childbirth Expectation/Experience Scale Version B | first 24 hours after birth
  The Wijma Childbirth Expectation/Experience Scale Version B (W-DEQ-B) was developed by Wijma et al. (1998) to measure the fear of childbirth experienced by women after childbirth. The scale consists of 32 items. Responses are numbered from 0 to 5 and are a six-point Likert-type scale. 0 represents "completely," and 5 represents "not at all." The minimum score on the scale is 0, while the maximum score is 160.
Depression Anxiety Stress Scale-21 | In the 28th week of pregnancy, After completing the program (4 weeks), 1st month postpartum, 3rd month postpartum
  The Depression Anxiety Stress Scale-21 was developed by Lovibond and Lovibond (1995), and its Turkish validity and reliability study was conducted by Sarıçam (2018). The scale consists of 21 items, with 7 items each in the depression, anxiety, and stress subscales. It assesses depression, anxiety, and stress symptoms in the past week on a four-point scale from (0) never to (3) always. A score of 5 or higher on the depression subscale, 4 or higher on the anxiety subscale, and 8 or higher on the stress subscale indicates a relevant problem.

CONTACTS AND LOCATIONS:
Locations (1):
- Ordu University, Ordu, Ordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Preventing Postpartum Depression With Mindful Self-Compassion Intervention A Randomized Control Study — https://journals.lww.com/jonmd/fulltext/2020/02000/preventing_postpartum_depression_with_mindful.3.aspx

DOCUMENTS (2):
  • Informed Consent Form: Intervention (2025-09-13): https://cdn.clinicaltrials.gov/large-docs/57/NCT07187557/ICF_001.pdf
  • Informed Consent Form: form (2025-09-13): https://cdn.clinicaltrials.gov/large-docs/57/NCT07187557/ICF_000.pdf